CLINICAL TRIAL: NCT05153057
Title: Longitudinal Cohort Study of Patients With Birdshot Chorioretinopathy.
Brief Title: Birdshot Chorioretinopathy : Prospective Follow-up and Immunogenetic Studies(CO-BIRD)
Acronym: CO-BIRD
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16002
Record Dates: First submitted 2021-01-12; First posted 2021-12-10 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Birdshot Chorioretinopathy; Posterior Uveitis
Keywords: Prospective follow-up; birdshot chorioretinopathy.
MeSH Terms: conditions — Birdshot Chorioretinopathy; Uveitis, Posterior | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted DNA Transformed cell lines from white cells Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Birdshot chorioretinopathy: Patients with a diagnosis of birdshot chorioretinopathy, with confirmed HLA-A29 positivity.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — The goal of the study is purely observational. Treatment decisions will be made by physicians according to the grading of the intraocular inflammation related to birdshot chorioretinopathy and to their consequences on visual function. These treatment decisions will be independent from the observational study.

SUMMARY:
The purpose of this study is twofold:

1. To analyze the clinical features of a cohort of patients with birdshot chorioretinopathy (BCR), an inflammatory bilateral ocular disease, affecting the choroid and the retina.

   Various imaging techniques will be used to assess the effect of the disease on the retina and the choroid.

   A standardized assessment of the visual function will be performed with visual acuity, visual field and color vision testing. The quality of life of the patients will be evaluated with the VFQ-25 questionnaire.

   These analyses will help delineating different forms of the disease among its heterogeneous presentations.
2. To identify predisposing factors for the disease. The condition is unique from the immunogenetic standpoint by its association with the HLA-A29 allele, which is the strongest link between an HLA class I antigen and a disease. To date, however, the mechanisms leading to birdshot chorioretinopathy remain unknown. GWAS (Genome Wide association Study) based on DNA of the cohort patients will be performed with the aim to identify other susceptibility genes associated with BCR.

DETAILED DESCRIPTION:
Birdshot chorioretinopathy is a bilateral chronic posterior uveitis that has been named in 1980. The "birdshot lesions" are the hallmark of the disease. In their most typical aspect these lesions are ovoid shaped hypopigmented spots at the level of the choroid.

One of the main difficulties of the diagnosis lies in the spectrum of presentations of the disease. The typical birdshot lesions are ovoid with their main axis oriented toward the optic disc. However, some are round and the can be clearly seen on fundus examination while others can be limited to subtle depigmentations. Typical lesions are one-quarter to one-half disc diameters, but confluent lesions may yield larger areas of depigmentation that are difficult to recognize. Although the typical lesions are depigmented, their presentation may change over time and pigment or atrophy may replace the initial cream-colored spots. The typical location, or the most easily seen location of the spots, is nasal to the optic disc. However, involvement of the posterior pole inside the temporal arcade is also possible. The spots usually predominate in the mid-periphery, but may also extend to the equator. A standardized classification of the birdshot lesions according to their size, their number, their pigmentation and their localization has been suggested to help in the categorization of the various disease presentations and for the longitudinal follow-up of affected patients. Spots clearly visible at the time of the diagnosis may disappear later. Hence, if the diagnosis of the birdshot chorioretinopathy is not made when spots are clearly visible, later presentations may not meet the definition commonly used for the disease. The disappearance of birdshot spots after treatment has been documented, but the effect of treatment on spots has not yet been assessed in large cohorts of patients. Indocyanine green angiography has been suggested as a reliable method to detect spots. However, it remains to be validated by a randomized assessment comparing indocyanine green angiography to color photographs for the detection of birdshot lesions.

Fluorescein angiography is useful in patients with birdshot chorioretinopathy to assess disease activity. In active disease, angiographic findings include leakage of the retinal veins, macular edema and optic disk hyperfluorescence. These findings are not disease specific, but they require a careful examination of the fundus seeking subtle spots when birdshot lesions are not obvious.

Given the above, the first goal of our prospective cohort study is to assess the heterogeneity of the disease, its spectrum of presentation and its evolution over time.

One of the characteristics of birdshot chorioretinopathy is its association with the HLA-A29 allele, which constitutes the strongest link between a disease and class I HLA allele. The mechanism by which HLA-A29 confers a risk for birdshot chorioretinopathy is a key question that remains unanswered. As with other associations between HLA class I antigens and diseases (HLA-B27 with spondylarthropathies and HLA B51 with Behçet's disease), the physiopathogeny of these links have not been elucidated.

Other factors playing a role in the physiopathogeny of the disease and not linked to the major histocompatibility complex are researched. A few families of patients with birdshot chorioretinopathy have been reported, which could point to additional genetic factors for disease susceptibility but does not rule out an environmental effect.

Hence, the complex physiopathology of birdshot chorioretinopathy could involve the HLA-A29 allele, other unknown genetic factors, as well as environmental factors.

Given the above, we are planning a GWAS (Genome Wide association Study) based on DNA of the cohort patients, which will be performed with the aim to identify other susceptibility genes associated with BCR.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral disease
2. Presence of at least three peripapillary "birdshot lesions" inferior or nasal to the optic disk in one eye
3. Low-grade anterior segment intraocular inflammation (defined as ≤ 1+cells in the anterior chamber)
4. Low grade vitreous inflammatory reaction (defined as ≤ 2+ vitreous haze‡) Supportive findings

1. HLA-A29 positivity 2. Retinal vasculitis 3. Cystoid macular edema

Exclusion Criteria:

1. Keratic precipitates
2. Posterior synechiae
3. Presence of infectious, neoplastic, or other inflammatory diseases that can cause multifocal choroidal lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the Department of Ophthalmology in a Paris University Hospital. Tertiary center for rare inflammatory ocular disorders.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2004-11-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Through study completion, an average of 1 year
  Standard decimal clarity for distance visual acuity. It is expressed from 0 which is minimum & worse value, corresponding to no light perception; to 1.0 (20/20) which is maximum & best value
Visual field testing | Through study completion, an average of 1 year
  Humphrey 30-2 automated threshold perimetry with foveal sensitivity. It is expressed in Mean Deviation from -25 decibels or unachievable which is minimum & worse value, to 0 decibel, which is maximum & best value.
Color vision | Through study completion, an average of 1 year
  Assessed with Desaturated Lanthony 15-Hue Test: an objective technic evaluating sensitivity to color & colour vision deficiency. Test result is categorized as Abnormal for minimum & worse evaluation; and Normal for maximum & best evaluation.
National Eye Institute 25-Item Visual Function Questionnaire | Through study completion, an average of 1 year
  Using a scale from 0 for minimum & worse, to 100 for maximum & best result; this questionnaire measures influence of visual impairment on various dimensions of quality of life such as emotional well-being and social functioning

SECONDARY OUTCOMES:
Assessment of birdshot spot size | Through study completion, an average of 1 year
  It describes appearance of the birdshot spots as small for minimum or large for maximum.
Assessment of birdshot spot number | Through study completion, an average of 1 year
  Spots are counted and categorized as <10 for minimum value & >50 for maximum
Assessment of birdshot spot localization | Through study completion, an average of 1 year
  Spots are categorized as Juxtapapillary, Equator & Diffuse.
Assessment of birdshot spot pigmentation | Through study completion, an average of 1 year
  Spot pigmentation is analysed and categorized as No pigmentation for minimum & Sever for maximum.
Assessment of edema | Through study completion, an average of 1 year
  Papillary & macular edema are analysed by Optical Coherence Tomography, using a scale from 0 to 4 respectively for minimum & best, to maximum & worse value.
Assessment of retinal vasculitis | Through study completion, an average of 1 year
  Arterial & venous vasculitis are analysed by Fluorescein Angiography, using a scale from 0 to 4 respectively for minimum & best, to maximum & worse value.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BREZIN, PhD & MD, Principal Investigator — Université de Paris, Ophtalmopôle, Hôpital Cochin, Assistance Publique - Hôpitaux de Paris.
Locations (1):
- Ophtalmopôle, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Sharing of anonymized clinical data with other investigators experienced in the care of patients with birdshot chorioretinopathy.

REFERENCES:
- [Background] Levinson RD, Brezin A, Rothova A, Accorinti M, Holland GN. Research criteria for the diagnosis of birdshot chorioretinopathy: results of an international consensus conference. Am J Ophthalmol. 2006 Jan;141(1):185-7. doi: 10.1016/j.ajo.2005.08.025. PMID 16386995
- [Background] Monnet D, Brezin AP, Holland GN, Yu F, Mahr A, Gordon LK, Levinson RD. Longitudinal cohort study of patients with birdshot chorioretinopathy. I. Baseline clinical characteristics. Am J Ophthalmol. 2006 Jan;141(1):135-42. doi: 10.1016/j.ajo.2005.08.067. PMID 16386987
- [Background] Monnet D, Brezin AP. Birdshot chorioretinopathy. Curr Opin Ophthalmol. 2006 Dec;17(6):545-50. doi: 10.1097/ICU.0b013e3280109479. PMID 17065923
- [Background] Holland GN, Shah KH, Monnet D, Brezin AP, Yu F, Nusinowitz S, Levinson RD. Longitudinal cohort study of patients with birdshot chorioretinopathy II: color vision at baseline. Am J Ophthalmol. 2006 Dec;142(6):1013-8. doi: 10.1016/j.ajo.2006.06.065. Epub 2006 Aug 2. PMID 17157585
- [Background] Monnet D, Levinson RD, Holland GN, Haddad L, Yu F, Brezin AP. Longitudinal cohort study of patients with birdshot chorioretinopathy. III. Macular imaging at baseline. Am J Ophthalmol. 2007 Dec;144(6):818-828. doi: 10.1016/j.ajo.2007.08.011. Epub 2007 Oct 18. PMID 17949671
- [Background] Gordon LK, Monnet D, Holland GN, Brezin AP, Yu F, Levinson RD. Longitudinal cohort study of patients with birdshot chorioretinopathy. IV. Visual field results at baseline. Am J Ophthalmol. 2007 Dec;144(6):829-837. doi: 10.1016/j.ajo.2007.08.010. Epub 2007 Oct 15. PMID 17937923
- [Background] Levinson RD, Du Z, Luo L, Monnet D, Tabary T, Brezin AP, Zhao L, Gjertson DW, Holland GN, Reed EF, Cohen JH, Rajalingam R. Combination of KIR and HLA gene variants augments the risk of developing birdshot chorioretinopathy in HLA-A*29-positive individuals. Genes Immun. 2008 Apr;9(3):249-58. doi: 10.1038/gene.2008.13. Epub 2008 Mar 13. PMID 18340360
- [Background] Kappel PJ, Monnet D, Yu F, Brezin AP, Levinson RD, Holland GN. Contrast sensitivity among patients with birdshot chorioretinopathy. Am J Ophthalmol. 2009 Feb;147(2):351-356.e2. doi: 10.1016/j.ajo.2008.08.021. Epub 2008 Oct 29. PMID 18973873
- [Background] Levinson RD, Monnet D, Yu F, Holland GN, Gutierrez P, Brezin AP. Longitudinal cohort study of patients with birdshot chorioretinopathy. V. Quality of life at baseline. Am J Ophthalmol. 2009 Feb;147(2):346-350.e2. doi: 10.1016/j.ajo.2008.08.011. Epub 2008 Oct 9. PMID 18848319
- [Background] Pagnoux C, Mahr A, Aouba A, Berezne A, Monnet D, Cohen P, Levinson RD, Brezin AP, Guillevin L. Extraocular manifestations of birdshot chorioretinopathy in 118 French patients. Presse Med. 2010 May;39(5):e97-e102. doi: 10.1016/j.lpm.2009.12.005. Epub 2010 Mar 10. PMID 20219319
- [Background] Brezin AP, Monnet D, Cohen JH, Levinson RD. HLA-A29 and birdshot chorioretinopathy. Ocul Immunol Inflamm. 2011 Dec;19(6):397-400. doi: 10.3109/09273948.2011.619295. PMID 22106906
- [Background] Dastiridou AI, Bousquet E, Kuehlewein L, Tepelus T, Monnet D, Salah S, Brezin A, Sadda SR. Choroidal Imaging with Swept-Source Optical Coherence Tomography in Patients with Birdshot Chorioretinopathy: Choroidal Reflectivity and Thickness. Ophthalmology. 2017 Aug;124(8):1186-1195. doi: 10.1016/j.ophtha.2017.03.047. Epub 2017 Apr 26. PMID 28456419
- [Background] Cunningham ET, Levinson RD, Denniston AK, Brezin AP, Zierhut M. Birdshot Chorioretinopathy. Ocul Immunol Inflamm. 2017 Oct;25(5):589-593. doi: 10.1080/09273948.2017.1400800. No abstract available. PMID 29144845
- [Background] Bousquet E, Khandelwal N, Seminel M, Mehanna C, Salah S, Eymard P, Bodin Hassani S, Monnet D, Brezin A, Agrawal R. Choroidal Structural Changes in Patients with Birdshot Chorioretinopathy. Ocul Immunol Inflamm. 2021 Feb 17;29(2):346-351. doi: 10.1080/09273948.2019.1681472. Epub 2019 Nov 12. PMID 31714872
- [Derived] Ferreira de Moura T, Enjalbert A, Monnet D, Kecili S, Imikerene L, Loeliger J, Thorne JE, Brezin AP. Peripapillary atrophy in patients with birdshot chorioretinitis. Br J Ophthalmol. 2025 Jul 22;109(8):882-887. doi: 10.1136/bjo-2024-326440. PMID 40010761
- [Derived] Kaisari E, Loeliger J, Thorne JE, Monnet D, Imikirene L, Kecili S, Brezin AP. Quality of Life in Patients with Birdshot Chorioretinitis Aged 80 and Older. Ocul Immunol Inflamm. 2025 Feb;33(2):280-286. doi: 10.1080/09273948.2024.2400172. Epub 2024 Sep 9. PMID 39250617
- [Derived] Debillon L, Thorne JE, Bousquet E, Duraffour P, Kecili S, Monnet D, Brezin AP. Birdshot Chorioretinitis in Patients Aged 80 and Older. Ocul Immunol Inflamm. 2024 Sep;32(7):1212-1217. doi: 10.1080/09273948.2023.2215322. Epub 2023 May 19. PMID 37204866